CLINICAL TRIAL: NCT00867256
Title: Large Diameter Metal-on-Metal Total Hip System IDE
Brief Title: Cormet Large Diameter Metal on Metal (LDMOM) Total Hip System (G030265)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated for business reasons; study closed.
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LDMOM
Record Dates: First submitted 2008-04-07; First posted 2009-03-23 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Avascular Necrosis
Keywords: arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Large Diameter Metal on Metal (Experimental)
  Interventions: Device: Large Diameter Metal on Metal

INTERVENTIONS:
Device: Large Diameter Metal on Metal

SUMMARY:
To demonstrate the safety and efficacy of the Cormet Large Diameter Metal on Metal (LDMOM) Total Hip System using a composite clinical success (CCS) primary endpoint.

DETAILED DESCRIPTION:
The results from the Cormet Large Diameter Metal on Metal (LDMOM) Total Hip System cohort will be compared to the historical results from a ceramic on ceramic (CoC) hip system cohort. The primary endpoint clinical composite success (CCS) criterion at 24 months postoperative is based on a Harris Hip Score ≥ 80 and the absence of any revision,replacement, or modification of any study component.

ELIGIBILITY:
INCLUSION CRITERIA:

Patient:

* is skeletally mature
* is mentally capable of completing follow-up forms
* will be available for follow-up out to 2 years
* has a preoperative Harris Hip Score <70 points
* has been deemed a candidate for hip replacement by diagnosis of the investigator.

EXCLUSION CRITERIA:

Patient:

* has active joint infection
* has had previous hip arthrodesis (fusion)
* has had above knee amputation of either extremity
* has active neoplastic disease
* has a need for a structural bone graft in the operative side
* has an ipsilateral hemi or total arthroplasty of any kind
* has a nonunion or malunion of any part of the femur on operative side
* has severe osteoporosis of the pelvis and/or femur as noted on standard radiograph
* is a prisoner
* is pregnant
* is known to be allergic to implant materials
* is morbidly obese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2004-03-31 (Actual); Primary Completion 2006-10-23 (Actual); Study Completion 2009-04-27 (Actual)

PRIMARY OUTCOMES:
Composite clinical criterion | 24-months postoperative
  Based on Harris Hip Score ≥ 80, and absence of any revision, replacement, or modification of any study component

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Carli, Study Director — Corin Ltd